CLINICAL TRIAL: NCT01124344
Title: Placebo-Controlled, Ascending Multiple-Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BMS-866949 in Healthy Subjects
Brief Title: Safety and Pharmacology Study of BMS-866949
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN166-002; 2010-018461-38 (EudraCT Number)
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Placebo or BMS-866949 (3 mg) (Active Comparator): Panel 1: Healthy Male Subjects
  Interventions: Drug: Placebo; Drug: BMS-866949
- Placebo or BMS-866949 (10 mg) (Active Comparator): Panel 2: Healthy Male Subjects
  Interventions: Drug: Placebo; Drug: BMS-866949
- Placebo or BMS-866949 (30 mg) (Active Comparator): Panel 3: Healthy Male Subjects
  Interventions: Drug: Placebo; Drug: BMS-866949
- Placebo or BMS-866949 (45 mg) (Active Comparator): Panel 4: Healthy Male Subjects
  Interventions: Drug: Placebo; Drug: BMS-866949
- Placebo or BMS-866949 (60 mg) (Active Comparator): Panel 5: Healthy Male Subjects
  Interventions: Drug: Placebo; Drug: BMS-866949
- Placebo or BMS-866949 (90 mg) (Active Comparator): Panel 6: Healthy Male Subjects
  Interventions: Drug: Placebo; Drug: BMS-866949
- Placebo or BMS-866949 (3 - 60 mg) (Active Comparator): Panel 7: Females
  Interventions: Drug: Placebo; Drug: BMS-866949

INTERVENTIONS:
Drug: Placebo — Oral Solution, Oral, 0 mg, Once Daily, 14 days
Drug: BMS-866949 — Oral Solution, Oral, 3 mg, Once Daily, 14 days
  Arms: Placebo or BMS-866949 (3 mg)
Drug: BMS-866949 — Oral Solution, Oral, 10 mg, Once Daily, 14 days
  Arms: Placebo or BMS-866949 (10 mg)
Drug: BMS-866949 — Oral Solution, Oral, 30 mg, Once Daily, 14 days
  Arms: Placebo or BMS-866949 (30 mg)
Drug: BMS-866949 — Oral Solution, Oral, 45 mg, Once Daily, 14 days
  Arms: Placebo or BMS-866949 (45 mg)
Drug: BMS-866949 — Oral Solution, Oral, 60 mg, Once Daily, 14 days
  Arms: Placebo or BMS-866949 (60 mg)
Drug: BMS-866949 — Oral Solution, Oral, 90 mg, Once Daily, 14 days
  Arms: Placebo or BMS-866949 (90 mg)
Drug: BMS-866949 — Oral Solution, Oral, 3-60 mg, Once Daily, 14 days
  Arms: Placebo or BMS-866949 (3 - 60 mg)

SUMMARY:
The main purpose of this study is to determine whether multiple doses.of BMS-886949 are safe and tolerable

ELIGIBILITY:
Inclusion Criteria:

* Panels 1-6: Healthy Male Subjects
* Panel 7: Females
* Ages 21 to 55, inclusive
* Body Mass Index (BMI) of 18 to 32 kg/m², inclusive
* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations

Exclusion Criteria:

* History of glaucoma or a confirmed intraocular pressure indicative of glaucoma at screening. (Normal IOP <21 mmHg)
* History or family history of psychiatric disorder
* Current treatment with prescription medication
* Exposure to any investigational drug or placebo within 12 weeks of study drug administration

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Assessment of safety by evaluating incidence of adverse events (AE) | Over a period of 28 days (+/- 2 days) of first dose

SECONDARY OUTCOMES:
Assessment of pharmacokinetics by evaluating plasma concentration versus time data | Over a period 28 days (+/- 2 days) of first dose
Assessment of pharmacodynamics by evaluating brain transporter occupancy | Over a period 28 days (+/- 2 days) of first dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Uppsala, Sweden

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx